CLINICAL TRIAL: NCT02225288
Title: A Study of E2022 Tape Formulation (Overlay-integrated E2022 18 mg Tape Formulation) for Different Application Sites and Intervals in Japanese Healthy Elderly Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2022-J081-007
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Subjects
Keywords: Healthy Subjects; Japanese; Males

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Period 1: Apply one E2022 tape to the designated site (back or upper arm) for 24 hours (applying in the morning and removing next morning) Period 2: Apply one E2022 tape to the designated site (back or upper arm, but different from Period 1) for 24 hours (applying in the morning and removing next morning) Period 3: Apply one E2022 tape to back (contralateral to Period 1 and 2). After the specified intervals (Group A: 48 hours), apply a new E2022 tape to the same site (for 24 hours after the first and second applications [applying in the morning and removing next morning])
  Interventions: Drug: E2022
- Group B (Experimental): Period 1: Apply one E2022 tape to the designated site (back or upper arm) for 24 hours (applying in the morning and removing next morning) Period 2: Apply one E2022 tape to the designated site (back or upper arm, but different from Period 1) for 24 hours (applying in the morning and removing next morning) Period 3: Apply one E2022 tape to back (contralateral to Period 1 and 2). After the specified intervals (Group B: 72 hours), apply a new E2022 tape to the same site (for 24 hours after the first and second applications [applying in the morning and removing next morning])
  Interventions: Drug: E2022
- Group C (Experimental): Period 1: Apply one E2022 tape to the designated site (back or chest) for 24 hours (applying in the morning and removing next morning) Period 2: Apply one E2022 tape to the designated site (back or chest, but different from Period 1) for 24 hours (applying in the morning and removing next morning) Period 3: Apply one E2022 tape to back (contralateral to Period 1 and 2). After the specified intervals (Group C: 96 hours), apply a new E2022 tape to the same site (for 24 hours after the first and second applications [applying in the morning and removing next morning])
  Interventions: Drug: E2022
- Group D (Experimental): Period 1: Apply one E2022 tape to the designated site (back or chest) for 24 hours (applying in the morning and removing next morning) Period 2: Apply one E2022 tape to the designated site (back or chest, but different from Period 1) for 24 hours (applying in the morning and removing next morning) Period 3: Apply one E2022 tape to back (contralateral to Period 1 and 2). After the specified intervals (Group D: 120 hours), apply a new E2022 tape to the same site (for 24 hours after the first and second applications [applying in the morning and removing next morning])
  Interventions: Drug: E2022

INTERVENTIONS:
Drug: E2022 — transdermal E2022 tape formulation (8.1 cm x 8.1 cm)

SUMMARY:
This is a single-center, 4-group, open-label study in Japanese healthy elderly males. A total of 48 subjects will be randomized to one of four groups (A to D, 12 subjects/group) to administer one E2022 tape to designated sites.

DETAILED DESCRIPTION:
This study consists of Screening, Treatment Period, and Follow-up. The Treatment Period is subdivided into three periods (Periods 1 to 3). Screening will start within 4 weeks before starting Treatment Period 1. In Treatment Periods 1 and 2, one E2022 tape will be applied to the designated site. The Treatment Period 2 application must have at least a 17-day interval from the end of Treatment Period 1 application. In Treatment Period 3, E2022 tape will be applied to back site (contralateral to the first applied site during Treatment Periods 1 and 2) after at least 17 days from the end of Treatment Period 2 (removing). A new E2022 tape will be applied to the same site after the specified intervals from the end of previous application (removing) in each group. Follow-up will start after at least a 17-day interval from the end of re-application in the Treatment Period 3 (removing).

ELIGIBILITY:
Inclusion Criteria

1. Male non-smokers (not smoking at least 4 weeks before Period 1) aged 65 years or older at informed consent
2. BMI at screening is 18.5 kg/m2 or above - below 28.0 kg/m2
3. Written informed consent
4. Given full explanation of this study and is willing to and able to comply with the protocol requirements

Exclusion Criteria

1. Have a current or past history of disorder requiring medical treatment within 8 weeks before the first application or infection within 4 weeks before the first application
2. Have a disorder within 4 weeks before the first application which affects the evaluation of study drug such as psychiatric, gastrointestinal, hepatic, renal, respiratory, endocrinological, hematological, neurological or cardiovascular system, or congenital metabolic abnormality
3. Have a history of gastrointestinal surgery (e.g., liver, kidney, digestive tract) which affects the pharmacokinetics of study drug
4. Have a history of treatment-requiring drug or food allergy or seasonal allergy at screening
5. Had caffeine-containing food or drink or alcohol within 72 hours before study drug application in Period 1
6. Had nutritional supplements, herbal preparations (including oriental medicines) or others (e.g., grapefruit-containing food or beverage) which may affect drug metabolizing enzymes and transporters, within 1 week before Period 1
7. Have used liquid products (including cosmetics) on study application sites (back, upper limb, chest), patch, tape or bandage, within 4 weeks before Period 1
8. Present or past clinical signs of skin hypersensitivity to topical product or atopic dermatitis
9. Excessively hairy or have shaved at application sites (back, upper limb, chest) within 4 weeks before Period 1
10. Eczema, dermatitis, abnormal pigmentation, injury, or scar at application sites which may affect the evaluation of skin symptoms

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number and frequency of adverse events | 168 hours after the end of application

SECONDARY OUTCOMES:
Pharmacokinetics of E2022: Cmax | 216 hours after the end of application
  Maximal Drug Concentration (Cmax)
Pharmacokinetics of E2022: AUC | 216 hours after the end of application
  Area Under the Plasma Concentration-Time Curve (AUC)
Pharmacokinetics of E2022: Tmax | 216 hours after the end of application
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Pharmacokinetics of E2022: t1/2 | 216 hours after the end of application
  Plasma Decay Half-Life (t1/2)

CONTACTS AND LOCATIONS:
Locations (1):
- Kagoshima, Kagoshima-ken, Japan